CLINICAL TRIAL: NCT01562093
Title: Effect of Intranasal Corticosteroids on Pulmonary Symptoms in Asthmatics With Nasal Congestion, a Randomized Controlled Trial
Brief Title: Effect of Intranasal Corticosteroids on Pulmonary Symptoms in Asthmatics With Nasal Congestion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational drugs no longer available
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/158
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Adrenal Cortex Hormones; Spirometry; Administration, Intranasal; Nasal blockage; Nasal sprays
MeSH Terms: conditions — Asthma; Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- local nasal steroids (Experimental)
  Interventions: Drug: corticosteroid nasal spray
- placebo (Placebo Comparator)
  Interventions: Drug: placebo nasal spray

INTERVENTIONS:
Drug: corticosteroid nasal spray — fluticasone furoate 55 µg (formula containing anhydrous glucose, dispersible cellulose, polysorbate 80, benzalkonium chloride, disodium edetate, purified water) once daily in each nostril for 3 months
  Other Names: Avamys
  Arms: local nasal steroids
Drug: placebo nasal spray — formula containing anhydrous glucose, dispersible cellulose, polysorbate 80, benzalkonium chloride, disodium edetate, and purified water, once daily in each nostril for 3 months
  Arms: placebo

SUMMARY:
In this study we will investigate the effect of intranasal corticosteroid therapy, which is known to reduce mucosal inflammation and nasal blockage, on asthmatic symptoms.

DETAILED DESCRIPTION:
Although up to 95% of asthma patients suffer from blocked nose, the majority of these patients do not undergo systematic assessment and treatment for nasal blockage. This is unfortunate, as optimal diagnosis and treatment of nasal blockage in asthmatics can reduce asthma morbidity and use of anti-asthmatic medication.

The "Unified Airways" concept considers the upper and lower airways as one unified airway. In recent years there has been increasing awareness about the relationship between inflammation in the upper and lower airways, with disease in the upper airways affecting the lungs through neurological, immunological and mechanical mechanisms, resulting in asthmatic symptoms.

Conditioning and filtration of the inspired air are important functions of the nose, and oral breathing results in inhalation of poorly conditioned and filtered air in to an already inflamed lower airway. Together will these mechanisms lead to a worsening of the asthmatic disease.

The aim of this study is to investigate the effect of intranasal corticosteroid therapy, which is known to reduce mucosal inflammation and nasal blockage, on asthmatic symptoms. The primary outcome variable is improvement in asthma symptomatology. The secondary outcome variables are improvement in nasal blockage.

ELIGIBILITY:
Inclusion Criteria:

* asthma (according to British Thoracic Society guideline)
* >18 years

Exclusion Criteria:

* pregnancy
* systemic disease with nasal manifestations
* cancer of the nose
* currently receiving cancer therapy
* previous nose surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume | up to 12 weeks
  spirometry, methacholine and mannitol

SECONDARY OUTCOMES:
improvement in nasal blockage | up to 12 weeks
  Sino-Nasal Outcome Test 20 (SNOT20), acoustic rhinometry (AR) and peak nasal inspiratory flow (PNIF)
nasal and exhaled NO | up to 12 weeks
  NO level in the nasal and exhaled air is measured by the chemiluminescence method with a LR 2000 nitric oxide gas analyser (Logan Research, Rochester, UK)
wheeze | up to 12 weeks
  Pulmotrack wheeze meter
subjective improvement in asthma symptomatology | up to 12 weeks
  Asthma Control Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Steinsvåg, MD prof, Study Director — St. Olav University Hospital, Trondheim, Norway; Malcolm Sue-Chu, MD, Principal Investigator — St Olavs University Hospital Trondheim; Vegard Bugten, MD, Principal Investigator — St Olavs University Hospital Trondheim
Locations (1):
- St Olav University Hospital, Trondheim, Norway